CLINICAL TRIAL: NCT06595472
Title: Effect of Plant Sterol-Enriched Palm Oil on Lipid Profile and Systemic Inflammation in Hyperlipidemic Adults: A Placebo-Controlled Double-Blinded Trial
Brief Title: Plant Sterol-Enriched Palm Oil to Improve Lipid Profile and Inflammation in Hyperlipidemic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pertanian Bogor (Other)
Collaborators: BASF (Industry)
Responsible Party: Principal Investigator, Mira Dewi, Dr, Assistant Professor, Principal Investigator, Head of Health and Nutrition Division at Seafast Center IPB, Institut Pertanian Bogor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-L/IPB/4202
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hyperlipidemias
Keywords: hyperlipidemia; plant sterol; C-reactive protein; Indonesia
MeSH Terms: conditions — Hyperlipidemias | interventions — Phytosterols; Palm Oil

STUDY DESIGN:
Intervention Model Description: The study was designed as a double-blinded randomized controlled trial, with 8 week intervention period, and conducted in Bogor district, West Java, Indonesia. The study subjects were volunteers residing in Bogor city and Bogor district, with known mild-moderate hypercholesterolemia. Subjects were supplied with either control or treatment cooking oil bottle every week, to be consumed as substitution of usually used cooking oil.
Who Masked: Participant, Investigator
Masking Description: The treatment and control cooking oil were indistinguishable in appearance and taste. The investigators and participants remained blinded to individual subject assignment throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plant sterol-enriched palm oil (Experimental): The group given cooking oil (palm oil) which is Enriched with Plant Sterol.
  Interventions: Dietary Supplement: Palm Oil Enriched with Plant Sterols
- palm oil (Placebo Comparator): The group given cooking oil (palm oil) which has the same composition and physical appearance as the intervention oil, but without plant sterol.
  Interventions: Dietary Supplement: Palm oil

INTERVENTIONS:
Dietary Supplement: Palm Oil Enriched with Plant Sterols — The enriched palm oil contained 52 mg/L of phytosterols, to reach the estimated intake of plant sterols in the treatment group at the level of around 2 g/day [22]. The phytosterols used was Vegapure 95 FF® derived from soybean derivatives containing campesterol, stigmasterol and beta-sitosterol. The oil is consumed by respondents as cooking oil.
  Arms: plant sterol-enriched palm oil
Dietary Supplement: Palm oil — The type, composition, and physical appearance of the oil is the same as those of the intervention arm, except that it was not added plant sterol. The oil is consumed by respondents as cooking oil.
  Arms: palm oil

SUMMARY:
This is a placebo-controlled double-blinded trial aimed to evaluate the effect of palm oil enriched with plant sterols on lipid profile and systemic inflammation marker in 100 adult hyperlipidemic residents of Bogor, Indonesia. Subjects were assigned to intervention oil which contained plant sterol and control oil which was the same as the intervention oil but did not contain plant sterol for 8 weeks. Data collected included nutritional status, energy and macronutrients consumption, blood lipid profile and inflammatory marker (hsCRP).

DETAILED DESCRIPTION:
Cardiovascular diseases, including coronary heart disease (CHD), are currently positioned amongst the leading causes of mortality globally. Risk factors of CHD include, among others, hypercholesterolemia and elevations in systemic inflammation. Functional foods enriched with compounds showing cholesterol-lowering effects are considered as one among various dietary and lifestyle intervention strategies to tackle this problem. A CHD-preventive effect of dietary plant sterols has been broadly discussed, not only due to their ability to reduce blood cholesterol level, but also to their proven anti-inflammatory potential. Palm oil is one amongst the most widely consumed edible oils in the world. Up to date, despite its widespread use, especially in Asian countries, no study has been conducted using palm oil as a vehicle for plant sterols. The aim of the placebo-controlled double-blinded trial presented here was therefore to evaluate the effect of palm oil enriched with plant sterols, used as a cooking oil, on lipid profile and systemic inflammation marker in 100 adult hyperlipidemic residents of Bogor, Indonesia. The study had 2 arms; intervention group in which subjects were given oil which contained plant sterol and control group which in which subjects were given the same oil as the intervention group but did not contain plant sterol for 8 weeks. The oil was consumed as cooking oil. Data on energy, macro nutrients, and cooking oil consumption were collected through interviews at baseline, week 2, 4, 6, and endline. Body weight and height measurement for nutritional status assessment and blood sample collection for biomarker analysis was conducted at baseline and endline.

ELIGIBILITY:
Inclusion Criteria:

* aged 25-60y
* total cholesterol concentration ≥200 mg/dL
* not requiring lipid-lowering drug therapy during the trial

Exclusion Criteria:

* secondary hyperlipidemia
* fasting triglyceride concentration >3.5 mmol/L
* body mass index >35 kg/m2
* use of any lipid-lowering drug
* suffering from gastrointestinal diseases or severe concomitant diseases

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Blood lipid profile | 8 weeks
  Concentration of blood HDL, LDL, triacylglycerols, and cholesterol (total) of participants after intervention period.

SECONDARY OUTCOMES:
Inflammatory marker | 8 weeks
  Concentration of high sensitivity C-Reactive protein of participants after intervention period.